CLINICAL TRIAL: NCT04129242
Title: Optimization of Closed-loop Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) as a Neurorehabilitation Tool
Brief Title: taVNS for Upper Limb Rehabilitation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Bashar Badran, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00086291; 5P20GM109040 (NIH)
Record Dates: First submitted 2019-09-23; First posted 2019-10-16 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Stroke
Keywords: Stroke; Rehabilitation; Vagus Nerve Stimulation; Brain Stimulation; Occupational Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "paired" taVNS + Task Specific Training (Active Comparator)
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) + Task Specifc Training
- "unpaired" taVNS + Task Specific Training (Active Comparator)
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) + Task Specifc Training

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) + Task Specifc Training — A closed-loop taVNS system that delivers taVNS with upper-limb rehabilitation training in a chronic stroke population.

SUMMARY:
This study explores the use of a new form of neuromodulation known as transcutaneous auricular vagus nerve stimulation (taVNS) which stimulates the ear. This stimulation will be delivered concurrently with upper limb motor rehabilitation training (3 days/week for 4 weeks) in chronic stroke patients. Patients will undergo a series of baseline assessments (including a brain scan), a 4-week course of motor rehabilitation, and post-assessments (including a second brain scan)

DETAILED DESCRIPTION:
This study aims to refine and develop closed loop taVNS, establish activity with key biomarkers, and show initial feasibility in a small clinical trial. For paired taVNS to succeed as a clinical treatment, it is critical to develop and refine a closed-loop taVNS platform that delivers stimulation concurrently during specific movements of the motor rehabilitation training.

Aim 1 develops this novel motion-gated closed-loop system that delivers taVNS in synchrony with specific upper limb motor activation (n=5) Aim 2 will combine the development of the closed-loop system with the investigator's mechanistic understanding to explore an open-label pilot trial (n=20) using closed-loop taVNS paired with task-specific training to determine the feasibility, safety, and potential effect size of this novel combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Ischemic or hemorrhagic stroke that occurred at least 6 months prior
* Completed conventional rehabilitation therapy at least one month prior
* Unilateral limb weakness with Fugl Meyer-Upper Extremity Scale score less than or equal to 58 (out of 66)

Exclusion Criteria:

* Primary intracerebral hematoma, or subarachnoid hemorrhage
* Bilateral upper extremity weakness
* Other concomitant neurological disorders affecting upper extremity motor function
* Documented history of dementia before or after stroke
* Documented history of uncontrolled depression or psychiatric disorder either before or after stroke which could affect their ability to participate in the experiment
* Uncontrolled hypertension despite treatment, specifically SBP (Systolic Blood Pressure) / DBP (Diastolic Blood Pressure) >=180/100mmHg at baseline
* Contraindicated for MRI scanning.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | "Paired" taVNS + Task Specific Training | "Unpaired" taVNS + Task Specific Training
Started | 10 | 10
Completed | 9 | 8
Not Completed | 1 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Adults with unilateral motor deficits post-stroke
Groups:
- Total: Total of all reporting groups
Arm/Group | "Paired" taVNS + Task Specific Training | "Unpaired" taVNS + Task Specific Training | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 5 | 13
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.33 (8.28) | 58.71 (6.45) | 57.93 (7.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Fugl-Meyer Assessment of the Upper Extremity
Description: The Fugl-Meyer Assessment of the Upper Extremity (FMA-UE) is a stroke rehabilitation assessment of arm/hand movement impairment. It is scored by assigning 30 items assessing voluntary arm/hand movements and 3 items assessing reflexes an ordinal rating (0=unable, 1=partial, 2=near normal), then summing the ratings to obtain a general statement of ability. Possible aggregate scores range from 0/66 to 66/66 points. Higher scores indicate greater levels of arm movement ability.
Time Frame: Mean change in FMA-UE score after 4 weeks of rehab, compared to baseline
Population: Adults with unilateral motor deficits post-stroke
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | "Paired" taVNS + Task Specific Training | "Unpaired" taVNS + Task Specific Training
Number analyzed (Participants) | 9 | 7
score on a scale | 5 (1.02) | 3.14 (0.63)

ADVERSE EVENTS:
Time Frame: 1 year, 8 months
Arm/Group | "Paired" taVNS + Task Specific Training | "Unpaired" taVNS + Task Specific Training
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT04129242/Prot_001.pdf
  • Informed Consent Form (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT04129242/ICF_002.pdf